CLINICAL TRIAL: NCT06220539
Title: CAsting and REhabilitation Versus Supervised Neglect for Osteochondral Lesions of the Talus in the Pediatric Population: The CARE Study, A Multicenter, Stratified, Block-Randomized Controlled Trial
Brief Title: CAsting and REhabilitation Versus Supervised Neglect for Osteochondral Lesions of the Talus in the Pediatric Population
Acronym: CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tristan Buck (Other)
Collaborators: Emma Childrens Hospital Foundation (Unknown); European Paediatric Orthopaedic Society (EPOS) (Unknown)
Responsible Party: Sponsor-Investigator, Tristan Buck, PhD candidate, MD, MSc, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL78874.018.22
Record Dates: First submitted 2023-05-25; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cartilage Injury; Orthopedic Disorder; Skeletal Injury; Rehabilitation; Physiotherapy
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Casting and Supervised Rehabilitation (Experimental): Patients in the intervention group will undergo non-weightbearing immobilization for 8 weeks in phase one: 4 in a circular cast with non-weightbearing followed by 4 weeks toe-tip weightbearing (10-20% of body weight) in a walking boot during daytime and a removable cast at night. In phase 2, a supervised rehabilitation will be performed till week 16 after which phase 3 will start at week 16-18
  Interventions: Other: Casting and supervised rehabilitation
- Standard Care (No Intervention): Patients in the control group will undergo the standard care. Standard care (''skill-full'' neglect) is described as adjustment of activities within the boundaries of pain. They can perform all activities wanted, except for painful activities. Patients and caretakers will be advised on the amount of activities by specialized orthopedic surgeons and periodical evaluation, and adjustment, will take place at the regular follow-up moments which is the same as in the intervention group. In this group, no supervised training or rehabilitation will be performed.

INTERVENTIONS:
Other: Casting and supervised rehabilitation — casting (8 weeks) followed by supervised rehabilitation
  Arms: Casting and Supervised Rehabilitation

SUMMARY:
Rationale: OCLs (osteochondral lesions) of the talus can be congenital or can occur after trauma or in patients with juvenile idiopathic arthritis (JIA). The main complaint of an OCL is pain during weightbearing activities. Therefore, these lesions have significant impact on the health status of patients.

Objective: The aim of this study is to optimize the treatment for skeletally immature patients with an osteochondral lesion. The hypothesis is that a period of immobilization and supervised rehabilitation will lead to better clinical and radiological outcomes compared with standard care which is a ''skill-full'' neglect.

Study design: Observational comparative study

Study population: Skeletally immature children with an osteochondral lesion of the talus diagnosed on CT.

Intervention: Patients in the intervention group will undergo an 8-week period of casting and walking on crutches. Afterwards, they will receive a protocolled period of rehabilitation under supervision of a physical therapist. The control group will have the standard care as treatment.

Main study parameters/endpoints: the main study outcome is the difference between the two groups on the OxAFQ-C. Secondary study outcomes are radiologic changes in terms of morphology and lesion size, NRS during weight bearing and quality of life measured with a Peds-QL, EQ-5D-y and AAS.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: the burden that patients will have is mainly the time that they have to spent on fulfilling the questionnaires.

DETAILED DESCRIPTION:
STUDY DESIGN After the diagnostic process in the outpatient clinics, patients will be counseled for both options, ''skill-full'' neglect or casting and supervised rehabilitation in a shared decision makig process. This process includes the choice talk, option talk, and decision talk. After the decision, patients will be placed in group one or two based on their preference.

Treatment groups Group 1: patients in the intervention group will undergo non-weightbearing immobilization for 8 weeks in phase one: 4 in a circular cast with non-weightbearing followed by 4 weeks toe-tip weightbearing (10-20% of body weight) in a walking boot during daytime and a removable cast at night. In phase 2, a supervised rehabilitation will be performed till week 16 after which phase 3 will start at week 16-18.

Group 2: Patients in the control group will undergo the standard care. Standard care (''skill-full'' neglect) is described as adjustment of activities within the boundaries of pain. They can perform all activities wanted, except for painful activities. Patients and caretakers will be advised on the amount of activities by specialized orthopedic surgeons and periodical evaluation, and adjustment, will take place at the regular follow-up moments which is the same as in the intervention group. In this group, no supervised training or rehabilitation will be performed.

STUDY POPULATION Population (base) All patients, up from June 2023, visiting the outpatient clinic of the orthopedic department in one of the participating hospitals will be screened for eligibility to participate in this study. Patients ≥4 years are considered as eligible as it is observed that OLTs can occur in this young population as well. In order to make the results of this study generalizable to this population and to optimize their treatment, it is decided to include this young patient group. If patients are eligible, they, and their caretakers will be informed about this study. After confirmation, patients will be allocated to one of the two groups. There are no restrictions on the number of inclusions per center.

Sample size calculation The sample size is calculated based on a minimally important difference of 17% in the OxAFQ-C physical domain. For this sample size calculation, a SD of 25 is used. A calculated sample size of 35 patients in each group is needed for an 80% study power. To compensate for potential loss to follow up of 7.5%, 38 patients will be included in both groups.

Main study parameter/endpoint The main study outcome is the difference in the end score of the OxAFQ-C questionnaire at 1-year follow-up.

Secondary study parameters/endpoints (if applicable) The secondary outcome is the cartilage repair during the radiologic follow up. Cartilage repair will be expressed in reduction of the lesion volume and surface.

Other study parameters (if applicable) The following baseline characteristics will be recorded: gender, age, body mass index, other musculoskeletal injuries, and level of sports pre-injury. Other important parameters of this study consist of the NRS weightbearing. The Peds-QL and EQ-5D-Y will be used to measure the quality of life of the participants. Returning to sport questions and AAS will be asked to compare return to sport outcomes and level of activity between the two groups.

Treatment allocation After the diagnostic process in the outpatient clinics, patients will be counseled for both options, ''skill-full'' neglect or casting and supervised rehabilitation in a shared decision makig process. This process includes the choice talk, option talk, and decision talk (11). After the decision, patients will be placed in group one or two based on their preference.

Study procedures Potential eligible patients will be screened before their initial presentation in our hospital based on the referral letter. At the initial presentation, patients will be seen at the outpatient clinic by the coordinating researcher and treating physician. In this consult they will be informed about the study. If needed, patients and care takers will have two working days to decide if they want to participate or not. After inclusion in the intervention (cast) group, patients will receive an appointment within one week to apply their cast.

The ankle function will be measured with the OxAFQ-C, which is a specific child tailored questionnaire (11). The NRS during weightbearing will be measured as this is a major complaint for patients suffering an osteochondral lesion of the talus. PedsQL and EQ-5D-youth will be measured for the monitoring of the quality of life.

Radiologic follow up will be as follows: patients will receive an X-ray at baseline in order to classify their skeletal maturity. MRI and CT scans will be conducted at baseline to provide a starting point in terms of radiologic characteristics. Furthermore, radiologic follow-up will be performed at 16 weeks, 1 year, 2 years, 5 years and 10 years after start of the treatment to detect the radiological change over time. However, the scans at baseline, one year and two years are considered as usual care, and the scans at 16 weeks, 5 years and 10 years will be for research aims.

Radiological characteristics that will be assessed at each radiologic follow up moment are as follows: lesion morphology, lesion size and bone marrow edema. Additionally, at the primary endpoint at 1 year, 2 blinded radiologists will measure each separately the above-mentioned radiologic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, osteochondral lesion of the talus
* Diagnosed on Computed Tomography (CT)
* Open physes of the distal tibia confirmed by a specialized musculoskeletal or pediatric radiologist
* Age ≥4 and ≤18

Exclusion Criteria:

* acute traumatic lesions
* surgically treated OLTs
* systemic diseases that can influence cartilage conditions (such as hemophilia)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Oxford Ankle Foot Questionnaire for Children (OxAFQ-C), physical domain | 1 year
  The response options to each item are on a 5-point scale rated from never (4), rarely (3), sometimes (2), very often (1) to always (0), where the number in brackets represents the value that should be applied by the scorer to each response. Domain scores are calculated as the total of the scale item scores divided by the maximum for each domain. Scores are ranged between 0-100. Higher scores represents better functioning.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) during weightbearing | 1 year
  pain severity during weightbearing using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
Pediatric Quality of Life Inventory | 1 year
  It is composed of 23 items that gauge function in the following four areas: physical (eight items), emotional (five items), social (five items), and school (five items). Patients report their function using a 5-point Likert scale ranging from 0 to 4. These responses are reverse scored and linearly transformed to a 0 to 100 scale, with a higher score indicating a higher QOL.
EuroQol Five Dimensions Health Questionnaire Youth (EQ5D-Y) | 1 year
  The EQ-5D-Y descriptive system comprises the following five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy. Each dimension has 3 levels: no problems, some problems and a lot of problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the younger patient's health state. This questionnaire reports the overall health of an individual on a 0% to 100% scale.
Return to Sport (level) | 1 year
  Lower-, same-, higher level than pre-injury
Return to Sport (time) | 1 year
  time in months
Radiological outcome (lesion morphology) | 1 year
  (change in) lesion morphology (cystic, crater, crater with fragment, crater with unstable fragment)
Radiological outcome (lesion size) | 1 year
  (change in) lesion size (surface in cm2 and volume in cm3)
Radiological outcome (bone marrow edema) | 1 year
  (change in) bone marrow edema (descriptive)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amphia Hospital Breda, Breda, Molengracht 21
  - Amsterdam UMC, Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided